CLINICAL TRIAL: NCT03580499
Title: A Pilot Study of the Effects of Vitamin B6 on Hot Flash Symptoms in Prostate Cancer Patients
Brief Title: Vitamin B6 in Reducing Hot Flashes in Participants With Prostate Cancer Undergoing Antiandrogen Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 18D.273; JT 12134 (Other: JeffTrial Number)
Record Dates: First submitted 2018-06-29; First posted 2018-07-09 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Hot Flashes; Prostate Carcinoma
MeSH Terms: conditions — Hot Flashes; Prostatic Neoplasms | interventions — Vitamin B 6

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive Care (vitamin B6) (Experimental): Participants receive vitamin B6 PO daily for 12 weeks.
  Interventions: Dietary Supplement: Vitamin B6; Other: Questionnaire Administration

INTERVENTIONS:
Dietary Supplement: Vitamin B6 — Given PO
  Other Names: 8059-24-3; VIT B6; Vitamin B-6; Vitamin B 6
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This pilot phase II trial studies how well vitamin B6 works in reducing hot flashes in participants with prostate cancer undergoing antiandrogen therapy. A nutritional supplement such as vitamin B6 may help improve hot flashes caused by antiandrogen therapy in participants with prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the effect of Vitamin B6 in improves the frequency or severity of hot flashes in prostate cancer patients receiving antiandrogen therapy (androgen deprivation therapy [ADT]).

OUTLINE:

Participants receive vitamin B6 orally (PO) daily for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are currently receiving ADT for prostate cancer and will continue on ADT for at least 13 weeks after enrollment. Patient may have been started on ADT at any past time point because patients experience hot flashes throughout ADT treatment
* Subjects are experiencing bothersome hot flashes per the study questionnaires
* Subjects are capable of giving informed consent.
* Willing to comply with all study procedures and be available for the duration of the study
* Able to obtain and take an acceptable form of vitamin B6

Exclusion Criteria:

* Subjects without a diagnosis of prostate cancer
* Subjects already receiving other treatment for hot flashes
* Subjects taking selective serotonin reuptake inhibitors (SSRIs)
* Subjects are currently taking vitamin supplementation which includes vitamin B6 at doses > 10 mg

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-09-13 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Median change in response to 10-point hot flash scale (1 = hot flash is not bothersome, 10 = hot flash is Most Severe) | Baseline to 8 weeks
  For the primary analysis, the difference in the median response to the 10-point hot flash scale between 8-week post-treatment and pre-treatment responses will be computed with the corresponding 95% percent confidence interval. The primary null hypothesis will be tested using a two-sided Wilcoxon Signed-Rank Test with alpha=0.05.

SECONDARY OUTCOMES:
Median change in response to 10-point hot flash scale (1 = hot flash is not bothersome, 10 = hot flash is Most Severe) | Baseline to 12 weeks
  The same approach will be used for the secondary analysis of 12-week post-treatment responses in comparison to the pre-treatment responses.

CONTACTS AND LOCATIONS:
Overall Officials: Costas Lallas, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/